CLINICAL TRIAL: NCT06178731
Title: Virtual Reality Reward Training and Transcranial Magnetic Stimulation for Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Peter Giacobbe, Psychiatrist, Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5159
Record Dates: First submitted 2023-12-01; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This is a non-blinded, randomized sham-controlled trial for effectiveness and feasibility of virtual reward reality training and rTMS for MDD with two arms. Patients with MDD who meet inclusion and exclusion criteria will be identified and recruited from the practices of Sunnybrook psychiatrists. Subjects will undergo either: i) VR RT + rTMS (n = 17) or ii) VR sham + rTMS (n = 17). Each treatment session involves: 12-15 min VR viewing, 15 min descriptive and imaginal recounting followed immediately by 3 min rTMS delivery with iTBS to the left DLPFC. The study will proceed according to the schedule laid out below. Both patients and treating team will be aware of all treatment parameters at all times.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality + rTMS (Experimental): Each treatment session involves: 12-15 min VR viewing, 15 min descriptive and imaginal recounting followed immediately by 3 min rTMS delivery with iTBS to the left DLPFC.
  Interventions: Device: rTMS; Other: Virtual Reality
- Virtual reality sham + rTMS (Sham Comparator): Each treatment session involves: 12-15 min VR viewing, 15 min descriptive and imaginal recounting followed immediately by 3 min rTMS delivery with iTBS to the left DLPFC.
  Interventions: Device: rTMS; Other: Virtual Reality

INTERVENTIONS:
Device: rTMS — 3 min rTMS delivery with iTBS to the left DLPFC
Other: Virtual Reality — 2-15 min VR viewing, 15 min descriptive and imaginal recounting

SUMMARY:
Anhedonia is a core feature of major depressive disorder (MDD) (DSM-5). Functional magnetic resonance imaging (fMRI) studies have associated anhedonia in MDD with altered frontostriatal activity and functional connectivity relative to controls. Conversely, antidepressant treatment is associated with increased ability for patients with MDD to sustain frontostriatal activity in a manner predictive of decrease in anhedonia and gains in daily positive affect. Novel interventions are needed to address anhedonia. Repetitive transcranial magnetic stimulation (rTMS) of the dorsolateral prefrontal cortex (DLPFC) has been shown to activate striatal reward circuits. Positive Affect Treatment (PAT) was developed to treat deficits in reward processing; a critical skill patients are trained on in PAT involves recounting and savouring of positive experiences. However, amotivation impedes some patients from engaging in positive activities, prompting the development of virtual reality reward training (VR RT) for this skill. Evidence is building that brain state at the time of rTMS impacts its therapeutic effect. For example, imaginal exposure and individualized symptom provocation just prior to rTMS enhances its therapeutic effect on post-traumatic stress disorder and obsessive-compulsive disorder, respectively. It is unknown whether VR RT can augment rTMS for MDD and if so whether it is mediated by enhancing changes in frontostriatal activity or functional connectivity.

The current study is significant for multiple reasons. As mentioned, there is a paucity of effective treatments for anhedonia and this study may inform development of a novel treatment strategy that harnesses findings from affective neuroscience. Recent economic analysis suggests that rTMS can be more cost-effective than pharmacotherapy or ECT for treatment-resistant depression (Ontario Health, 2021). Our findings will provide insight on ways to synergize specific psychotherapeutic techniques with targeted stimulation of brain circuits to more effectively treat subtypes of depression.

DETAILED DESCRIPTION:
This is a non-blinded, randomized sham-controlled trial for effectiveness and feasibility of virtual reward reality training and rTMS for MDD with two arms. Patients with MDD who meet inclusion and exclusion criteria will be identified and recruited from the practices of Sunnybrook psychiatrists. Subjects will undergo either: i) VR RT + rTMS (n = 17) or ii) VR sham + rTMS (n = 17). Each treatment session involves: 12-15 min VR viewing, 15 min descriptive and imaginal recounting followed immediately by 3 min rTMS delivery with iTBS to the left DLPFC. The study will proceed according to the schedule laid out below. Both patients and treating team will be aware of all treatment parameters at all times.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female or male patients between ages 18-65 2. Diagnosis of major depressive disorder as defined by the Diagnostic and Statistical Manual fifth edition (DSM-5) 3. Hamilton Rating Scale for Depression (17-item) score of at least 16 4. Clinically significant anhedonia as defined by a Smith-Hamilton Pleasure Scale (SHAPS) score of at least 20 (Krystal et al., 2020) 5. On a stable antidepressant regimen for at least 4 weeks before treatment which can continue during treatment and agreement to not make changes or additions to psychotropic medications during the course of their participation in the study 6. Ability to provide informed consent and comply with all testing, follow-ups and study appointments and protocols

Exclusion criteria:

1. Any past or current evidence of psychosis or mania
2. Active neurologic disease
3. Any lifetime history of seizures
4. Alcohol or substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
5. Current active suicidal ideation
6. Personality disorder deemed to be the primary pathology
7. Taking more than 2 mg lorazepam (or an equivalent) or any anticonvulsant
8. Previous rTMS treatment
9. Lifetime history of non-response to an adequate course (minimum 8 treatments) of electroconvulsive therapy
10. Previous or current engagement in ketamine treatment for major depressive disorder
11. Any contraindication to MRI scanning
12. Likely to relocate or move out of the country during the study's duration (3-4 months from baseline visit)
13. Frequent motion sickness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-10-29 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
The Hamilton Depression Rating Scale | up to 4 weeks after treatment
  Mood symptoms, higher scores mean worse outcome. Min = 0, Max = 52

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada